CLINICAL TRIAL: NCT05645276
Title: A Phase Ia/Ib, Open Label, Dose Escalation and Dose Extension Trial of Anti-PD-1 and LAG-3 Bispecific Antibody AK129 to Evaluate the Safety, Tolerability and Antitumor Efficacy in Patients With Advanced Malignant Tumors
Brief Title: A Study of AK129 in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK129-101
Record Dates: First submitted 2022-11-17; First posted 2022-12-09 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Advanced Malignant Tumors(Stage IA-IB)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The dose escalation stage, pharmacodynamic confirmation stage and dose expansion stage of AK129 (Experimental): 7 dose groups were set up, which were 0.03mg/kg,0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg, 10 mg/kg and 25 mg/kg in dose escalation stage; 2-3 dose levels that do not exceed maximum tolerated dose(MTD) may be selected for pharmacodynamic confirmation cohort extension in pharmacodynamic confirmation stage;Five cohorts with different indications were included in each group with 10-20 subjects in dose expansion stage.
  Interventions: Drug: AK129 IV infusion

INTERVENTIONS:
Drug: AK129 IV infusion — AK129 is administered intravenously according to the frequency and dosage of administration at different stages.

SUMMARY:
A Phase Ia/Ib, open label, dose escalation and dose extension trial of Anti-PD-1 and LAG-3 bispecific antibody, AK129, to evaluate the safety, tolerability and antitumor efficacy in patients with advanced malignant tumors

DETAILED DESCRIPTION:
Anti Lymphocyte Activation Gene-3(LAG-3) combination therapy showed a preliminary antitumor signal in multiple solid tumors and hematologic tumor.LAG-3 targeted drug Relatilimab in a Phase 2/3 study comparing a combination of relatilimab and nivolumab to nivolumab alone in previously untreated patients with metastatic or unresectable melanoma.The combination therapy of Relatilimab with nivolumab showed a statistically significant and clinically significant progression-free survival(PFS) benefit compared to the nivolumab group, Because of this study, the FDA approved the combination therapy for first-line therapy of melanoma.

AK129 is a humanized immunoglobulin G1(IgG1) bispecial antibody(BsAb), which can bind anti-programmed death receptor 1(PD-1) and LAG-3 at the same time, and block the interaction of PD-1/programmed cell death - ligand 1(PD-L1), LAG-3/ major histo-compatibility complex II(MHCII),etc. The aim of the first human, dose-escalation study of this investigational drug is to explore its safety, tolerability, and initial antitumor efficacy, and to evaluate its pharmacokinetic and pharmacokinetic characteristics to identify the appropriate dose and regimen.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the written informed consent form(ICF) voluntarily.
2. Aged ≥ 18 to ≤ 75 years.
3. Eastern Cooperative Oncology Group(ECOG) performance status score of 0 or 1.
4. Life expectancy≥ 3 months.
5. Histologically or cytologically confirmed advanced solid tumors(dose-escalation phase) or selected tumor species(pharmacodynamic confirmation phase and dose-expansion phase);Patients with advanced metastatic malignancies who have failed first-line, or second-line, or third-line, or fourth-line standard therapy, or are ineligible for standard therapy, or cannot tolerate chemotherapy, or are unwilling to receive chemotherapy, or have no effective standard therapy.
6. Pharmacodynamic confirmation phase and dose expansion phase: at least one measurable tumor lesion(RECIST v1.1, lymphoma according to Lugano 2014 evaluation criteria).A lesion from a site previously treated with radiotherapy or other local regional therapy is considered a non-target lesion unless there is definite progression of the lesion or the neoplastic nature of the lesion is confirmed by biopsy.
7. Pharmacodynamic confirmation phase and dose extension phase: All subjects agree to provide archived or freshly obtained tumor tissue samples within 2 years prior to initial administration(formalin-fixed paraffin-embedded (FFPE) tissue wax blocks or approximately 10 unstained tumor tissue sections,and if there is archived tumor tissue within 6 months or 3 months, or freshly obtained tumor tissue, preferably recently obtained tumor tissue samples).
8. The results of laboratory examination during the screening period indicate that the subjects have good organ function:1).Hematology (no supportive treatment of any component blood and cell growth factors were used within 7 days prior to the start of the study):Neutrophil absolute value(ANC)≥1.5×10^9/L(solid tumors) or 1.0×10^9/L(lymphoma);Platelet count≥100×10^9/L(solid tumors) or 75×10^9/L(lymphoma);haemoglobin≥90 g/L or ≥5.6 mmol/L. 2).Kidney:Serum creatinine(Cr)≤1.5×Upper limit of normal(ULN),or Creatinine clearance *(CrCl) calculated value≥ 50 mL/min,CrCl was calculated by Cockcroft-Gault formula:CrCl (mL/min)={(140-age)×weight(kg)×F}/(SCr (mg/dL)×72),Male F=1,Female F=0.85,SCr=serum creatinine.3).Liver:Serum total bilirubin(TBil)≤1.5×ULN,Subjects with confirmed/suspected Gilbert disease,TBil ≤ 3× ULN;aspartate aminotransferase(AST) and alanine aminotransferase(ALT) ≤ 2.5×ULN,For subjects with liver metastasis or liver cancer,AST and ALT ≤ 5×ULN.4).Blood clotting function:Internationally standardized ratio(INR)≤ 1.5×ULN and activated partial thromboplastin time(APTT)≤ 1.5×ULN(If the subject is receiving anticoagulant therapy, the subject will receive a steady dose of anticoagulant and the coagulation parameters(prothrombin time(PT)/INR and APTT) will be within the expected range of anticoagulant therapy at the time of screening).5).Cardiac function:Left ventricular ejection fraction(LVEF)≥ 50%;Troponin protein T or I<2×ULN.
9. Fertile female subjects must undergo a negative serum pregnancy test within 3 days prior to initial medication.If a fertile female subject has sex with an unsterilized male partner, the subject must initiate a highly effective contraceptive method from screening and must agree to continue using these precautions until 120 days after the final administration of the study drug;Periodic abstinence, safe period contraception and extracorporeal ejaculation are not acceptable contraceptive methods;
10. If an unsterilized male subject has sex with a fertile female partner, the subject must use an effective contraceptive method from the beginning of screening to within 120 days after the last dose.

Exclusion Criteria:

1. Active central nervous system metastasis.
2. Subjects with uncontrolled pleural effusion, pericardial effusion, or abdominal effusion requiring repeated drainage(frequency greater than monthly).
3. Patients with other active malignant tumors within 2 years prior to the first administration, except for locally curable tumor species and those who have been cured, such as squamous cell carcinoma of the skin, basal cell carcinoma of the skin, superficial bladder carcinoma, and carcinoma in situ of the breast.
4. Known primary or secondary immunodeficiency,including human immunodeficiency virus(HIV) antibodies tested positive.
5. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
6. Known interstitial lung disease or non-infectious pneumonia requiring glucocorticoid therapy;Except for those caused by radiation therapy.
7. Severe infections, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia, occur within 4 weeks prior to initial administration.
8. Present with active infections(including active tuberculosis and active treponema pallidum) requiring systemic treatment, and have used systemic antibacterial, antiviral or antifungal drugs within 2 weeks prior to initial administration;Note: Antiviral drugs for viral hepatitis B are excluded.
9. Subjects with active viral hepatitis B, non-active or asymptomatic hepatitis B virus(HBV) carriers(Hepatitis B surface antigen(HBsAg) positive) with HBV deoxyribonucleic acid(DNA)>200IU/mL, and subjects with active viral hepatitis C.
10. Have active or documented inflammatory bowel disease(e.g. Crohn's disease, ulcerative colitis), active diverticulitis.
11. Any of the following cardiovascular and cerebrovascular diseases:a.Myocardial infarction, unstable angina pectoris, pulmonary embolism, aortic dissection, deep vein thrombosis, and any arterial thromboembolism events occurred within 6 months prior to initial administration;b.New York Heart Association(NYHA) cardiac functional grade ≥ II for heart failure;c. Severe arrhythmias requiring long-term drug intervention; Subjects with asymptomatic and stable ventricular frequency of atrial fibrillation were admitted.d.Uncontrolled hypertension(defined as systolic blood pressure>150 mmHg and diastolic blood pressure>100 mmHg) with sufficient antihypertensive medication, or a history of hypertensive crisis or hypertensive encephalopathy.
12. Received the following antitumor drugs or treatments before initial administration:a. Received monoclonal antibody drugs(including PD-1/L1) immunotherapy drugs within 6 weeks prior to initial administration or within 5 half-time period of the drug, whichever is shorter;b. Received small-molecule targeted drugs, immunomodulatory drugs , Chinese generic drugs with anti-tumor indications, or palliative radiotherapy within 2 weeks prior to initial administration;c. Received other types of antitumor therapy, including chemotherapy, radical radiotherapy, or any unapproved investigational drug within 4 weeks prior to initial dosing;d. Major surgical treatment within 4 weeks prior to initial administration.
13. Dose expansion phase: Immunocheckpoint inhibitors targeting LAG-3 were previously used.
14. Subjects requiring therapy with glucocorticoids(prednisone>10 mg/ day or equivalent of glucocorticoids) or other immunosuppressive agents within 14 days prior to initial administration;The following are excluded:a. Glucocorticoids as prophylactic drugs for hypersensitivity reactions(such as medication before Computed Tomography(CT) examination).
15. Live vaccine was administered within 4 weeks prior to initial administration.
16. No remission of toxicity from previous antitumor therapy was defined as failure to return to National Cancer Institute Common Terminology Criteria for Adverse Events(NCI CTCAE) v5.0≤1 or the level specified in the inclusion/exclusion criteria(except hair loss).
17. A known history of severe hypersensitivity to other monoclonal antibodies.
18. Any condition that the investigator believes may result in a risk of receiving the study drug or interfere with the evaluation of the study drug or the subject's safety or the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events(AE) | Up to approximately 2 years
  Incidence and severity of AEs is aim to evaluate the safety of AK129
Incidence of serious adverse events(SAE) | Up to approximately 2 years
  Incidence of SAE is aim to evaluate the safety of AK129
The incidence of suspected unexpected serious adverse reactions(SUSAR) | Up to approximately 2 years
  The incidence of SUSAR is aim to evaluate the safety of AK129
Incidence of dose-limiting toxicity(DLT) | Up to approximately 2 years
  The purpose of DLT is to find the Phase II recommended dose(RP2D) or MTD
Number of participants with clinically significant changes in laboratory assessment data as assessed by CTCAE v5.0. | Up to approximately 2 years
  Monitor and summerize all data derive from clinically significant changes in laboratory assessment data per Common Terminology Criteria for Adverse Events(CTCAE)5.0.
AE that leads to the termination or suspension of treatment | Up to approximately 2 years
  AE that leads to the termination or suspension of treatment is aim to evaluate the safety of AK129

SECONDARY OUTCOMES:
Objective response rate(ORR) | Up to approximately 2 years
  ORR is proportion of subjects with complete response(CR) or partial response(PR), based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1(Solid Tumor)or Lugano 2014 Evaluation Criteria(lymphoma)
Disease control rate(DCR) | Up to approximately 2 years
  Disease control rate(DCR) is defined as the proportion of subjects achieving a best of response(BOR) of confirmed CR and PR and stable disease(SD) per RECIST v1.1(Solid Tumor)or Lugano 2014 Evaluation Criteria(lymphoma)
duration of response(DoR) | Up to approximately 2 years
  Duration of response(DoR) is defined as the period from the first documentation of confirmed response(CR or PR) to the first documentation of progressive disease(PD) (as per RECIST v1.1(Solid Tumor)or Lugano 2014 Evaluation Criteria(lymphoma)) or death due to any cause, whichever occurs first
time to response(TTR) | Up to approximately 2 years
  Time to response(TTR) is defined as the time from the first dose of investigational products until the first confirmation of CR or PR
progression-free survival(PFS) | Up to approximately 2 years
  Progression-free survival(PFS) is defined as the time from the first dose of investigational products until documentation of PD(progressive disease)(as per RECIST v1.1) or death due to any cause, whichever occurs first.
overall survival(OS) | Up to approximately 2 years
  Overall survival(OS) is defined as the time from the first dose of investigational products until death due to any cause.
The drug concentration of AK129 in serum | Up to approximately 2 years
  The drug concentration of AK129 in serum was used to assess the blood concentration of AK129 at different dosing time points.
maximum concentration(Cmax) | Up to approximately 2 years
  Maximum concentration(Cmax) is to evaluate the Pharmacokinetics(PK) of AK129.
peak time(Tmax) | Up to approximately 2 years
  Peak time(Tmax)is to evaluate the Pharmacokinetics(PK) of AK129.
half time(t1/2) | Up to approximately 2 years
  Half time(t1/2) is to evaluate the Pharmacokinetics(PK) of AK129.
area under curve(AUC) | Up to approximately 2 years
  Area under curve(AUC) is to evaluate the Pharmacokinetics(PK) of AK129.
clearance rate(CL) | Up to approximately 2 years
  Clearance rate(CL) is to evaluate the Pharmacokinetics(PK) of AK129.
apparent volume of distribution(Vd) | Up to approximately 2 years
  Apparent volume of distribution(Vd) is to evaluate the Pharmacokinetics(PK) of AK129.
Number and percentage of subjects with anti-drug antibody(ADA) to AK129 | Up to approximately 2 years
  The immunogenicity of AK129 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, Doctor, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No